CLINICAL TRIAL: NCT04749147
Title: Color Priming and Patient Decision-Making in the Emergency Department: Priming "Threat" in Patients With Low-Risk Chest Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHRISTUS Health (Other)
Responsible Party: Principal Investigator, Matthew Vandermause, DO, Principal Investigator, CHRISTUS Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2018-108
Record Dates: First submitted 2021-01-30; First posted 2021-02-11 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Chest Pain; Cardiac Event
Keywords: Emergency Department; HEART score
MeSH Terms: conditions — Chest Pain; Cardiovascular Diseases; Emergencies

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Black and White Print (Experimental): The survey concerns the patients' chest pain, perception of their safety, and their comfort with their discharge. This group's survey will be printed in black and white and feature black and white graphics.
  Interventions: Other: Black and White Printed Survey
- Red Print (Experimental): The survey concerns the patients' chest pain, perception of their safety, and their comfort with their discharge. This group's survey will be printed in red text and feature red graphics.
  Interventions: Other: Red Printed Survey

INTERVENTIONS:
Other: Black and White Printed Survey — This survey will feature black and white text and graphics.
  Arms: Black and White Print
Other: Red Printed Survey — This survey will feature red text and graphics.
  Arms: Red Print

SUMMARY:
This will be a prospective cross-sectional study evaluating a convenience sample of patients in the ED with low-risk chest pain defined by a HEART score of 3 or less.

DETAILED DESCRIPTION:
This will be a prospective cross-sectional study. We will evaluate a convenience sample of patients in the ED with low-risk chest pain defined by a HEART score of 3 or less. Patients will be consented for participation and will fill out one of two surveys concerning their chest pain and chances of adverse cardiac events based on their HEART score. One survey will be printed in red text and feature red graphics; the other will be printed in black-and-white and feature black and-white graphics. The surveys will otherwise be identical. Enrolled patients will be asked to fill out survey questions related to their perception of their safety and their comfort with their discharge.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years or age and older presenting to the ED with a complaint of chest pain who are found to have a HEART score of 3 or less.

Exclusion Criteria:

* Patients who refuse to provide consent.
* Patients unable to fill out the survey due to clinical instability, severe pain, or disorientation as determined by an emergency physician.
* Incarcerated patients.
* Patients who have a HEART score of >3.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Chest Pain Questionnaire | 2 years
  To assess a patient's level of relief/worry with being discharged from the emergency department (ED) after presenting with a chief complaint of chest pain and subsequently being informed they have a less than 2% chance of a major adverse cardiac event (heart attack) in the next six weeks. The questionnaire grades their level of relief/worry from (1) Very Relieved, (2) Somewhat Relieved (3) No Change (4) Somewhat Worried (5) Very Worried.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Vandermause, DO, Principal Investigator — CHRISTUS Health
Locations (1):
- CHRISTUS Health Spohn, Corpus Christi, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigator is interested in pursuing potential collaborations and grants in the future.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] The population studied will be a convenience sample of adult patients presenting to the ED with chest pain as a primary complaint who then are risk-stratified with the HEART score and are found to have a score of 3 or less.
- [Background] Gerend, Mary, and Sias, Tricia.
- [Background] majic, A., Merritt, S., Banister, C., and Blinebry, A. (2014).
- [Background] Shi J, Zhang C, Jiang F. Does red undermine individuals' intellectual performance? A test in China. Int J Psychol. 2015 Feb;50(1):81-4. doi: 10.1002/ijop.12076. Epub 2014 May 5. PMID 25611931
- [Background] Mehta R, Zhu RJ. Blue or red? Exploring the effect of color on cognitive task performances. Science. 2009 Feb 27;323(5918):1226-9. doi: 10.1126/science.1169144. Epub 2009 Feb 5. PMID 19197022
- [Background] Lutfey KE, Eva KW, Gerstenberger E, Link CL, McKinlay JB. Physician cognitive processing as a source of diagnostic and treatment disparities in coronary heart disease: results of a factorial priming experiment. J Health Soc Behav. 2010 Mar;51(1):16-29. doi: 10.1177/0022146509361193. PMID 20420292
- [Background] Gorini A, Pravettoni G. An overview on cognitive aspects implicated in medical decisions. Eur J Intern Med. 2011 Dec;22(6):547-53. doi: 10.1016/j.ejim.2011.06.008. Epub 2011 Jul 7. PMID 22075278
- [Background] Blumenthal-Barby JS, Krieger H. Cognitive biases and heuristics in medical decision making: a critical review using a systematic search strategy. Med Decis Making. 2015 May;35(4):539-57. doi: 10.1177/0272989X14547740. Epub 2014 Aug 21. PMID 25145577
- [Background] Elwyn G, Frosch D, Thomson R, Joseph-Williams N, Lloyd A, Kinnersley P, Cording E, Tomson D, Dodd C, Rollnick S, Edwards A, Barry M. Shared decision making: a model for clinical practice. J Gen Intern Med. 2012 Oct;27(10):1361-7. doi: 10.1007/s11606-012-2077-6. Epub 2012 May 23. PMID 22618581
- [Background] Stacey D, Bennett CL, Barry MJ, Col NF, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Legare F, Thomson R. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD001431. doi: 10.1002/14651858.CD001431.pub3. PMID 21975733
- [Background] Isaacs CG, Kistler C, Hunold KM, Pereira GF, Buchbinder M, Weaver MA, McLean SA, Platts-Mills TF. Shared decision-making in the selection of outpatient analgesics for older individuals in the emergency department. J Am Geriatr Soc. 2013 May;61(5):793-8. doi: 10.1111/jgs.12207. Epub 2013 Apr 16. PMID 23590177
- [Background] Hess EP, Knoedler MA, Shah ND, Kline JA, Breslin M, Branda ME, Pencille LJ, Asplin BR, Nestler DM, Sadosty AT, Stiell IG, Ting HH, Montori VM. The chest pain choice decision aid: a randomized trial. Circ Cardiovasc Qual Outcomes. 2012 May;5(3):251-9. doi: 10.1161/CIRCOUTCOMES.111.964791. Epub 2012 Apr 10. PMID 22496116
- [Background] Hess EP, Hollander JE, Schaffer JT, Kline JA, Torres CA, Diercks DB, Jones R, Owen KP, Meisel ZF, Demers M, Leblanc A, Shah ND, Inselman J, Herrin J, Castaneda-Guarderas A, Montori VM. Shared decision making in patients with low risk chest pain: prospective randomized pragmatic trial. BMJ. 2016 Dec 5;355:i6165. doi: 10.1136/bmj.i6165. PMID 27919865
- [Background] Chen JC, Cooper RJ, Lopez-O'Sullivan A, Schriger DL. Measuring patient tolerance for future adverse events in low-risk emergency department chest pain patients. Ann Emerg Med. 2014 Aug;64(2):127-36, 136.e1-3. doi: 10.1016/j.annemergmed.2013.12.025. Epub 2014 Feb 13. PMID 24530111
- [Background] Six AJ, Backus BE, Kelder JC. Chest pain in the emergency room: value of the HEART score. Neth Heart J. 2008 Jun;16(6):191-6. doi: 10.1007/BF03086144. PMID 18665203
- [Background] Backus BE, Six AJ, Kelder JC, Bosschaert MA, Mast EG, Mosterd A, Veldkamp RF, Wardeh AJ, Tio R, Braam R, Monnink SH, van Tooren R, Mast TP, van den Akker F, Cramer MJ, Poldervaart JM, Hoes AW, Doevendans PA. A prospective validation of the HEART score for chest pain patients at the emergency department. Int J Cardiol. 2013 Oct 3;168(3):2153-8. doi: 10.1016/j.ijcard.2013.01.255. Epub 2013 Mar 7. PMID 23465250